CLINICAL TRIAL: NCT00812994
Title: Blood Levels of Neurosteroids and Neurotrophic Factors in Normal Controls and in Patients With Major Depression
Brief Title: Neurotrophic Factors and Depression
Acronym: Lex/BDNF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Owen Wolkowitz, UCSF
Masking: Double | Purpose: Basic Science
Other Study IDs: H3097-19671-08
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Depression
Keywords: Depression; BDNF; neurotrophic factor; neurosetroid; allopregnanolone
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Escitalopram (Experimental)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — SSRI antidepressant
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study intended to determine if there are baseline differences in serum neurosteroid levels and neurotrophic factor (BDNF) levels in healthy controls vs unmedicated depressed subjects, and whether the levels of these change with antidepressant treatment. Study also intended to determine if baseline neurosteroid/ BDNF levels, and the change in these levels with =treatment, are correlated with clinical antidepressant response to escitalopram (Lexapro).

DETAILED DESCRIPTION:
The study was approved by the UCSF Committee on Human Research, and all participants gave informed consent. The depressed subjects began treatment with placebo for one week, followed by escitalopram for eight weeks (10 mg per day x 4 weeks, followed by 20 mg per day x 4 weeks, as tolerated) in a double-blind, fixed-order, within-subject cross-over manner. The depressed subjects and the psychiatric rater were unaware of the study design and the sequence and duration of treatments. Depressed and control subjects underwent venipuncture to obtain blood for assays. The controls underwent venipuncture once, and the depressed subjects had venipuncture just prior to beginning active escitalopram treatment and again after 8 weeks of escitalopram treatment. Blood was also collected at Weeks 4 and 8 of treatment in the depressed subjects for assay of citalopram and citalopram metabolites, to gauge medication compliance. Finally, depression severity and global clinical change were assessed in the depressed subjects at Baseline and at the end of Week 8 of escitalopram treatment.

ELIGIBILITY:
Male subjects with unipolar Major Depressive Disorder (DSM-IV) with a minimum score of 22 on the 10-item Montgomery-Åsberg Depression Rating Scale (MADRS) who were medication-free for at least 6 weeks, were enrolled. Fifteen individually age-matched (+ 3 years) healthy male controls with no history of psychiatric illness were also enrolled. Subjects' ages ranged from 22- 55 y.o. (mean + S.D.= 41.4 + 8.75 y.o.). All subjects were required to pass a urine toxicology screen (assessing the presence of drugs of abuse) on the day of testing.

Exclusion Criteria:

Individuals with co-morbid panic disorder were excluded, since they may poorly tolerate typical starting doses of antidepressants , and individuals with co-morbid post-traumatic stress disorder were excluded, since they may have neuroendocrine regulatory responses different from those of depressed subjects without PTSD. Exclusion criteria for both groups included recent (within 6 months) alcohol or drug abuse as defined by DSM-IV criteria, concurrent psychotherapeutic interventions, poor medical health or abnormal clinical labs, active suicidality, and use of medications that could interfere with the study.

Ages: 22 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Serum BDNF levels | Baseline, week 4, week 8
Serum allopregnanolone levels | Baseline, week 4, week 8

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | baseline, week 4, week 8
Clinical Global Impression | Baseline, week 4, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Owen M Wolkowitz, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - UCSF, San Francisco, California